CLINICAL TRIAL: NCT05701709
Title: An Open-Label, Single-Arm, Multi-Center Phase I Clinical Study to Evaluate the Safety, Tolerability, Efficacy and Pharmacokinetics of SHR-A2102 in Patients With Advanced Solid Tumors
Brief Title: Phase I Study of SHR-A2102 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A2102-I-102
Record Dates: First submitted 2023-01-18; First posted 2023-01-27 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-03

CONDITIONS: Advanced Solid Tumors

STUDY DESIGN:
Intervention Model Description: SHR-A2102 single arm
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHR-A2102 (Experimental)
  Interventions: Drug: SHR-A2102

INTERVENTIONS:
Drug: SHR-A2102 — SHR-A2102 was given intravenously. Patients may continue to use SHR-A2102 until disease progression or unacceptable toxicity occurs.

SUMMARY:
The study was designed to evaluate the efficacy, safety, and pharmacokinetics of SHR2102 in patients with advanced solid tumors. The objective of this study was to determine the dose-limiting toxicity, maximum tolerance and recommended dose of SHR-A2102 in phase II study.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent;
2. Age ≥18 years old, gender unlimited;
3. The physical status score of the Eastern Tumor Cooperative Group (ECOG) was 0 ~ 1;
4. Life expectancy Predicted survival ≥3 months;
5. Histologically or cytologically confirmed advanced or metastatic malignant tumor; Patients with advanced solid tumors confirmed by pathology who have failed or been intolerant to standard treatment, have no standard treatment or refuse standard treatment;
6. There is at least one measurable lesion that meets the RECIST 1.1 criteria.

Exclusion Criteria:

1. Plan to receive any other antitumor therapy during this trial;
2. Receiving other investigational drugs or treatments that are not on the market within 4 weeks prior to the initial administration of the study drug;
3. Received antitumor therapy such as chemotherapy, radiotherapy, biotherapy, targeted therapy, or immunotherapy within 4 weeks prior to first administration of the study drug (nitrosourea or mitomycin C within 6 weeks prior to first administration; Oral fluorouracil within 2 weeks prior to initial first administration); Palliative radiotherapy or local therapy within 2 weeks before first administration use of the study drug;
4. Had major surgery other than diagnosis or biopsy within 4 weeks prior to the study's initial dosing;
5. Treatment with CYP3A4, CYP2D6, P-gp or BCRP booster or inducer is less than 5 drug half-life from the date of first administration;
6. According to NCI-CTCAE v5.0, adverse events caused by previous antitumor therapy did not recover to ≤ grade 1 (except hair loss; In the judgment of the investigator, after consultation with the sponsor, some tolerable chronic grade 2 toxicity may be excluded);
7. Inadequately treated central nervous system (CNS) metastases, or the presence of uncontrolled or symptomatic active CNS metastases, may be characterized by the presence of clinical symptoms, cerebral edema, spinal cord compression, cancerous meningitis, pia meningeal disease, and/or rapid progression. Patients with CNS metastases that have been adequately treated and whose neurological symptoms return to baseline at least 4 weeks prior to randomization (except for residual signs or symptoms associated with CNS treatment) may be enrolled. In addition, subjects must either stop corticosteroids or receive prednisone (or an equivalent dose of another corticosteroid) at least 4 weeks prior to randomization;
8. Any other malignancies, excluding cured basal cell carcinoma of the skin and carcinoma in situ of the cervix, etc. within 5 years prior to initial administration;
9. A history of clinically significant lung disease (such as interstitial pneumonia, radiation pneumonia, pulmonary fibrosis) or chest imaging during screening suggests any such disease;
10. Severe infections that require intravenous antibiotic, antiviral or antifungal control;
11. Active HBV or HCV infection (HBsAg positive and viral copy number ≥2000 IU/mL, HCV antibody positive and HCV RNA higher than the lower limit of detection method);
12. History of immunodeficiency (including HIV positive, other acquired or congenital immunodeficiency diseases) or organ transplantation;
13. Concomitant diseases (such as severe diabetes, thyroid disease, and psychosis) or any other conditions that, in the investigator's judgment, seriously endanger the patient's safety or affect the patient's ability to complete the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 395 (Estimated)
Dates: Start 2023-04-06 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | 24 months
  Adverse events are assessed by CTCAE v5.0
Maximum tolerated dose (MTD) | 12 weeks
  MTD is defined as the maximum dose within the first 3 weeks of multiple dosing that does not exceed the proportion of subjects who develop DLT as specified in the protocol's BOIN design.
Recommended Phase 2 dose (RP2D) | 24 months
  RP2D will be determined based on the available data for toxicity and PK.
Dose Limiting Toxicity (DLT) | 3 weeks
  Adverse events that occurred during the DLT observation period (the first period of study administration, a total of 21 days) that were determined to be related to the study drug (see protocol for details).

SECONDARY OUTCOMES:
Peak plasma concentration (Cmax) | 12 weeks
Area under the plasma concentration versus time curve (AUC） | 12 weeks
T1/2 (Half-life) | 12 weeks
  The time required for the plasma concentration of a drug to be reduced by 50%
Immunogenicity: Number of subjects with anti-SHR-A2102 antibody (ADA), incidence, occurrence time, duration, etc | 12 weeks
Objective response rate (ORR) | 24 months
duration of response (DoR) | 24 months
disease control rate (DCR) | 24 months
progression-free survival (PFS) | 24 months
overall survival (OS) | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Chest Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided